CLINICAL TRIAL: NCT00424242
Title: A Pharmacokinetic Study of Pemetrexed in the Cerebrospinal Fluid of Patients With Leptomeningeal Metastases
Brief Title: Pemetrexed Disodium in the Cerebrospinal Fluid of Patients With Leptomeningeal Metastases
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 06C2; STU00004482 (Other: Northwestern University IRB)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Metastatic Cancer; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous Condition; Secondary Myelofibrosis; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; tumors metastatic to brain; leptomeningeal metastases; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; previously treated myelodysplastic syndromes; secondary acute myeloid leukemia; acute undifferentiated leukemia; mast cell leukemia; recurrent adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; T-cell large granular lymphocyte leukemia; atypical chronic myeloid leukemia, BCR-ABL negative; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; chronic myelomonocytic leukemia; refractory hairy cell leukemia; prolymphocytic leukemia; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; adult grade III lymphomatoid granulomatosis; intraocular lymphoma; post-transplant lymphoproliferative disorder; refractory multiple myeloma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; Waldenstrom macroglobulinemia; stage IV adult Burkitt lymphoma; recurrent adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; adult nasal type extranodal NK/T-cell lymphoma; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; secondary myelofibrosis; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; recurrent adult grade III lymphomatoid granulomatosis; stage III multiple myeloma; primary systemic amyloidosis; extramedullary plasmacytoma; monoclonal gammopathy of undetermined significance; isolated plasmacytoma of bone
MeSH Terms: conditions — Central Nervous System Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Neoplasm Metastasis; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Brain Neoplasms; Meningeal Carcinomatosis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, Mast-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Large Granular Lymphocytic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Intraocular Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Extranodal NK-T-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Immunoglobulin Light-chain Amyloidosis; Monoclonal Gammopathy of Undetermined Significance | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escalating doses of Pemetrexed (Experimental): Escalating doses of Pemetrexed beginning at 500 mg/m2
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Orally beginning at 500 mg/m2 every 3 weeks until disease progression
  Other Names: Alimta; LY231514

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Studying samples of cerebrospinal fluid and blood from patients with cancer in the laboratory may help doctors learn how pemetrexed disodium works in the body and identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying the side effects and how well pemetrexed disodium works in treating patients with leptomeningeal metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the cerebrospinal fluid (CSF):plasma ratio of pemetrexed disodium at different IV dose levels in patients with leptomeningeal metastases.
* Determine the safety of this drug in these patients.
* Determine the antitumor activity of this drug in these patients.
* Assess the role of CSF vascular endothelial growth factor and YKL 40 as markers of response and/or prognosis in these patients.

OUTLINE: Patients receive pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo lumbar puncture and blood collection prior to therapy and 30-60 minutes after the first dose of pemetrexed disodium for pharmacological studies. Patients with Ommaya reservoirs undergo cerebrospinal fluid (CSF) collection at baseline and 0.25, 0.50, 1, 2, 4, 6 and 8.0 hours after pemetrexed disodium administration. CSF is then obtained once during each subsequent course of study treatment. CSF and blood are also evaluated for YKL 40 and vascular endothelial growth factor.

After completion of study therapy, patients are followed every 2-3 months.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of systemic malignancy (solid tumor or hematologic malignancy) or primary CNS lymphoma with leptomeningeal metastases (LM) as documented by MRI, cerebrospinal fluid, or both
* Patients may have brain metastases in addition to LM
* Patients with clinically significant interstitial fluid with effusion controlled by drainage are eligible

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 2 months
* Creatinine clearance ≥ 45 mL/min
* Bilirubin < 1.5 times upper limit of normal (ULN)
* Transaminases < 3.0 times ULN (5 times ULN for hepatic metastasis)
* WBC > 3,000/mm³
* Neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 10 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Able to undergo lumbar puncture (i.e., no noncommunicating hydrocephalus or spinal block) or has an Ommaya reservoir in place
* Able to take steroids, cyanocobalamin (vitamin B12), and folic acid
* No other active cancer except nonmelanoma skin cancer or carcinoma in situ of the cervix
* Patients with prior malignancies who are in complete remission and are off all therapy for that malignancy for ≥ 3 years are eligible
* No significant medical or psychiatric illness that would interfere with study compliance

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* No nonsteroidal anti-inflammatory drugs (NSAIDs) or acetylsalicylic acid within 2 days before or after study treatment (5 days for long-acting NSAIDs)
* No other concurrent cytotoxic chemotherapy
* Concurrent hormonal or biological therapy allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Correlation of cerebrospinal fluid levels with plasma levels of different doses of pemetrexed disodium | Every 6 weeks for assessment while on study.
  Patients will have CSF collected approximately every 6 weeks for assessment while on study.
To determine whether there is any anti-tumor activity against LM with Pemetrexed. | Every six weeks.
  Patients will have a scan every six weeks to assess tumor response.
To determine the safety of Pemetrexed in patients with LM. | After every 2 doses approximately 6 weeks
  Adverse events will be collected every six weeks during patient visits.
To assess the role of serum biomarkers in patients with LM. | Prior to dose one
  Patients will have a one time blood draw to look at serum biomarkers prior to dose one.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States